CLINICAL TRIAL: NCT06935630
Title: Comparison of The Effect of 5-MTHF and Folic Acid Supplementation in Increasing Red Blood Cell Folate in Pregnant Women : A Randomized Controlled Trial Study
Brief Title: Comparison of The Effect of 5-MTHF and Folic Acid Supplementation in Increasing Red Blood Cell Folate in Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Prodia Diacro Laboratories P.T. (Industry); Simex Pharmaceutical Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Interventional
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pregnant Women
Keywords: Interventional; Folic Acid; Pregnant Women
MeSH Terms: interventions — Folic Acid; 5-methyltetrahydrofolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The folic acid supplementation codes will be blinded (double-blind) until all study phases are completed. This ensures that the participants, investigators, and outcomes assessors are unaware of which intervention each participant is receiving during the study. This helps to minimize potential bias in the evaluation of the treatment outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Folic Acid Group (Active Comparator): This group will receive daily oral supplementation of 600 mcg (1.35 μmol) of folic acid film-coated tablets for a duration of three months. Participants will be instructed to consume the supplement at a consistent time each day. Monitoring for compliance and potential side effects will be conducted throughout the study period
  Interventions: Dietary Supplement: Folic Acid
- 5-MTHF Group (Experimental): This group will receive daily oral supplementation of 1100 mcg (1.35 μmol) of 5-MTHF glucosamine salt (HY-FOLIC®) film-coated tablets for a duration of three months. Participants will be instructed to consume the supplement at a consistent time each day. Monitoring for compliance and potential side effects will be conducted throughout the study period.
  Interventions: Dietary Supplement: 5-MTHF (5-methyltetrahydrofolate)

INTERVENTIONS:
Dietary Supplement: Folic Acid — Participants in this group will receive a daily oral dose of 600 mcg (1.35 μmol) of folic acid in film-coated tablet form for a duration of three months. This synthetic form of folate will be administered to assess its impact on red blood cell folate levels compared to 5-MTHF.
  Other Names: Folic Acid 600 mcg (1.35 μmol)
  Arms: Folic Acid Group
Dietary Supplement: 5-MTHF (5-methyltetrahydrofolate) — Participants in this group will receive a daily oral dose of 1100 mcg (1.35 μmol) of 5-methyltetrahydrofolate (5-MTHF) glucosamine salt, specifically HY-FOLIC®, in film-coated tablet form for a duration of three months. This active form of folate will be administered to assess its impact on red blood cell folate levels compared to folic acid
  Other Names: HY-FOLIC® 1100 mcg
  Arms: 5-MTHF Group

SUMMARY:
This randomized controlled trial aims to compare the efficacy of 5-methyltetrahydrofolate (5-MTHF) and folic acid supplementation in increasing red blood cell (RBC) folate levels in pregnant women.

This study will recruit pregnant women and randomly assign them to receive either 5-MTHF or folic acid supplementation. The primary outcome is the difference in RBC folate levels between the two groups at the end of the study. Secondary outcomes include the proportion of women achieving a target RBC folate level of 906 nM, changes in plasma 5-MTHF, homocysteine, and unmetabolized folic acid (UMFA) levels from baseline to month three (M3).

The findings of this study will provide valuable insights into the comparative effectiveness of 5-MTHF and folic acid supplementation in optimizing folate status during pregnancy, potentially informing clinical practice and guidelines. All participants will be provided with detailed information about the study, and their participation will be voluntary. Ethical considerations, including informed consent and data confidentiality, will be strictly adhered to throughout the study.

DETAILED DESCRIPTION:
This prospective, double-blind, randomized controlled trial (RCT) aims to evaluate and compare the efficacy of 5-methyltetrahydrofolate (5-MTHF) and folic acid supplementation in increasing red blood cell (RBC) folate levels among pregnant women in their first trimester. The study is grounded in the understanding that both food folate and folic acid are metabolized into 5-MTHF, the active form of folate essential for DNA synthesis and homocysteine remethylation. Given the established links between folate deficiency, hyperhomocysteinemia, and adverse pregnancy outcomes, including neural tube defects (NTDs), pre-eclampsia, and premature birth, this research seeks to determine if 5-MTHF, as the direct active form, offers superior benefits over traditional folic acid supplementation. The findings will provide crucial insights into optimizing folate supplementation strategies during early pregnancy, potentially improving maternal and fetal health outcomes.

The study will recruit 100 pregnant women aged 25-35 years, with gestational ages between 9-14 weeks, who meet the inclusion criteria of normal BMI (18.5-24.9 kg/m2), hemoglobin levels above 11 g/dL, and a declaration of good health based on prior medical examinations. Participants will be randomly assigned to one of two groups: one receiving 600 mcg (1.35 μmol) of folic acid and the other receiving 1100 mcg (1.35 μmol) of 5-MTHF glucosamine salt (HY-FOLIC®), ensuring an equimolar dosage comparison. Exclusion criteria include pre-existing upper gastrointestinal diseases, history or current use of drugs interacting with folate metabolism (e.g., methotrexate), antiepileptic therapy, or concomitant use of proton pump inhibitors (PPIs), antacids, or H2 receptor blockers within the past three months. This rigorous selection process aims to minimize confounding variables and ensure the internal validity of the study.

The primary outcome of this research is to determine the difference in RBC folate levels between the two supplementation groups at the end of the three-month study period. Secondary outcomes include the proportion of pregnant women in each group achieving an RBC folate level threshold of 906 nM, as well as changes in plasma 5-MTHF, homocysteine, and unmetabolized folic acid (UMFA) levels from baseline to the end of the intervention period. These outcomes will provide a comprehensive assessment of the comparative effectiveness of 5-MTHF and folic acid in improving folate status and related biomarkers in pregnant women. Blood samples will be collected at baseline and at the end of the third month to measure these parameters, ensuring objective and quantifiable data for analysis.

Ethical considerations are paramount in this study. All participants will provide written informed consent prior to enrollment, and the study protocol will be reviewed and approved by an Institutional Review Board (IRB) or equivalent ethics committee. Participant confidentiality will be maintained throughout the study, and data will be anonymized during analysis and reporting. Any potential risks associated with blood sampling or supplementation will be thoroughly explained to participants, and appropriate safety measures will be implemented. Participants will be informed of their right to withdraw from the study at any time without penalty.

The results of this study are expected to contribute significantly to the current understanding of optimal folate supplementation during pregnancy, potentially impacting clinical guidelines and practices. By comparing 5-MTHF and folic acid directly, this research will provide evidence-based recommendations for healthcare providers to ensure adequate folate levels in pregnant women, thereby reducing the risk of adverse pregnancy outcomes and promoting maternal and fetal health.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a gestational age of 9-14 weeks
* Age: 25 - 35 years old
* Have normal BMI (18.5-24.9 kg/m2)
* Declared healthy based on previous health examinations
* Hb > 11 g/dl

Exclusion Criteria:

* Pregnant women with upper gastrointestinal disease
* History or current use of drugs interacting with folate metabolism (e.g., Methotrexate)
* History or current use of antiepileptic therapy
* Concomitant use of Proton Pump Inhibitors (PPI), antacid, and AH2 receptor blocker

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Red Blood Cell (RBC) Folate Levels | Baseline and Month 3 (End of Intervention)
  This measure will assess the difference in RBC folate levels between the 5-MTHF and folic acid supplementation groups. Blood samples will be collected at baseline and at the end of the 3-month intervention period. RBC folate levels will be quantified using a validated laboratory assay to determine the impact of each supplement on folate status. The red blood cell folate (RBC folate) levels in pregnant women who receive 5-MTHF supplementation expected to be higher than those who receive folic acid supplementation.

SECONDARY OUTCOMES:
Proportion of Participants Achieving Target RBC Folate Level | Month 3 (End of Intervention)
  The proportion of pregnant women in each supplementation group who achieve an RBC folate level of 906 nM at the end of the 3-month intervention period will be determined. This measure will assess the effectiveness of each supplement in reaching a clinically relevant threshold for folate status.
Change in Plasma 5-MTHF Levels | Baseline and Month 3 (End of Intervention)
  The change in plasma 5-MTHF levels from baseline to the end of the 3-month intervention period will be measured. This will assess the direct impact of each supplement on circulating 5-MTHF concentrations. The plasma 5-MTHF levels in pregnant women who receive 5-MTHF supplementation expected to be higher than those who receive folic acid supplementation.
Change in Plasma Homocysteine Levels | Baseline and Month 3 (End of Intervention)
  The change in plasma homocysteine levels from baseline to the end of the 3-month intervention period will be measured. This will assess the effect of each supplement on homocysteine metabolism, a key indicator of folate function. The serum homocysteine levels in pregnant women who receive 5- MTHF supplementation expected to be lower than those who receive folic acid supplementation.
Change in Plasma UMFA Levels | Baseline and Month 3 (End of Intervention)
  The change in plasma unmetabolized folic acid (UMFA) levels from baseline to the end of the 3-month intervention period will be measured. This will assess the accumulation of unmetabolized folic acid, providing insight into the metabolic handling of each supplement. The levels of Unmetabolized Folic Acid (UMFA) in pregnant women who receive 5-MTHF supplementation expected to be lower than those who receive folic acid supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Ernawati Ernawati, Doctor, Principal Investigator — Soetomo General Hospital Surabaya
Locations (1):
- Mulyorejo Public Health, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, we are undecided regarding the sharing of Individual Participant Data (IPD) from this study with other researchers. Several factors are currently under consideration, including the potential benefits of data sharing for advancing scientific knowledge, as well as the ethical and logistical challenges associated with ensuring participant privacy and data security. We are also evaluating the requirements and guidelines of potential data repositories and funding agencies. A final decision will be made after careful deliberation and consultation with relevant stakeholders, including the Institutional Review Board (IRB) or ethics committee, and will be documented accordingly